CLINICAL TRIAL: NCT04623216
Title: A Phase Ib/II, Open Label Study of Sabatolimab as a Treatment for Patients With Acute Myeloid Leukemia and Presence of Measurable Residual Disease After Allogeneic Stem Cell Transplantation
Brief Title: Sabatolimab as a Treatment for Patients With Acute Myeloid Leukemia and Presence of Measurable Residual Disease After Allogeneic Stem Cell Transplantation.
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Study was stopped following a strategic decision from the Sponsor. It was not based on any safety findings or safety concerns with sabatolimab.
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CMBG453F12201; 2020-000869-17 (EudraCT Number)
Record Dates: First submitted 2020-11-03; First posted 2020-11-10 (Actual); Results first posted 2025-06-03 (Actual); Last update posted 2025-10-16 (Actual); Status verified 2025-10

CONDITIONS: Acute Myeloid Leukemia
Keywords: Sabatolimab; MBG453; TIM-3; Azacitidine; Acute Myeloid Leukemia; AML; Allogeneic Hematopoietic Stem Cell Transplantation; aHSCT; Measurable Residual Disease; MRD; Phase Ib/II; Acute myeloid leukemia Hematopoietic stem cell transplantation
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Neoplasm, Residual | interventions — sabatolimab; Azacitidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Sabatolimab 400mg (Experimental): Safety cohort 1: Participants in this arm will receive sabatolimab 400mg intravenously every 4 weeks.
  Interventions: Biological: Sabatolimab
- Sabatolimab 800mg (Experimental): Safety cohort 2: Participants in this arm will receive sabatolimab 800mg intravenously every 4 weeks.
  Interventions: Biological: Sabatolimab
- Sabatolimab + Azacitidine (Experimental): Expansion cohort 3: Participants in this arm will receive sabatolimab at the recommended dose for expansion in combination with azacitidine.
  Interventions: Biological: Sabatolimab; Drug: Azacitidine
- Sabatolimab (Experimental): Expansion cohort 4: Participants in this arm will receive sabatolimab at the recommended dose for expansion.
  Interventions: Biological: Sabatolimab
- Sabatolimab (adolescent cohort) (Experimental): Adolescent safety cohort (cohort 5): ≥12 to < 18 year old adolescent participants in this arm will receive sabatolimab at the recommended dose for expansion.
  Interventions: Biological: Sabatolimab

INTERVENTIONS:
Biological: Sabatolimab — Sabatolimab is a solution in vial for IV infusion
  Other Names: MBG453
Drug: Azacitidine — Azacitidine comes in Vial for IV infusion or subcutaneous administration
  Arms: Sabatolimab + Azacitidine

SUMMARY:
The primary purpose of this study was to test the hypothesis that preemptive treatment with sabatolimab, alone or in combination with azacitidine, when administered to participants with Acute myeloid leukemia (AML)/secondary AML who were in complete remission with positive measurable residual disease post-allogeneic hematopoietic stem cell transplantation (Minimal residual disease (MRD)+ post- Allogeneic hematopoietic stem cell transplantation (aHSCT)), could enhance the graft versus leukemia (GvL) response and prevent or delay hematologic relapse without an unacceptable level of treatment-emergent toxicities, including clinically significant acute and/or chronic graft-versus-host disease (GvHD) and immune-related adverse events

DETAILED DESCRIPTION:
This is a phase Ib/II, open label, multi-center study of sabatolimab as monotherapy and in combination with azacitidine, in participants with AML/secondary AML who had received one aHSCT and achieved complete remission but MRD+, by local assessment, anytime at >= Day 60 after aHSCT and at least 2 weeks after immunosuppressive medications had been tapered off.

The study was planned to enroll approximately 59 participants and be conducted in two parts:

Part 1 was a Safety Run-in of approximately 20 participants, to assess whether sabatolimab as monotherapy at the two tested dose levels (400 mg and 800 mg intravenously Q4W) was safe when administered in the post-aHSCT setting. For each dose level, once the required number of evaluable participants had been confirmed, enrollment would be halted until participants had completed the dose limiting toxicities (DLT) observation period (≥ 8 weeks following the first dose). Following the observation period for DLTs, a Safety Review Meeting was to be conducted after each dose level to assess safety and determine the recommended dose for expansion to proceed with enrollment of additional cohorts in Part 2 of the study.

Part 2 consisted of sabatolimab monotherapy expansion cohort of approximately 13 participants, sabatolimab in combination with azacitidine cohort of approximately 20 participants, and an adolescent cohort of approximately 6 participants (≥ 12 years but < 18 years of age) with sabatolimab as monotherapy. Sabatolimab was to be administered at the recommended dose for expansion determined in Part 1.

After initiating Part 2, Novartis took the decision to put enrollment in permanent halt and terminate the sabatolimab program. This decision was not driven by any safety concerns.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent must be obtained prior to participation in the study.
* At the date of signing the informed consent form (ICF), eligible participants must be ≥ 18 years for the adult cohorts; and ≥ 12 years old but < 18 years old for the adolescent cohort (cohort 5), which will open after completion of Safety Run-in.
* Participants in complete remission (< 5% bone marrow blasts, absence of circulating blasts, and absence of extramedullary disease) with MRD positivity by local assessment or by central assessment where required (e.g., USA sites), any time at ≥ Day 60 after aHSCT
* Diagnosis of AML/secondary AML and received one prior aHSCT performed to control AML
* Ability to provide a fresh bone marrow aspirate sample collected within 28 days from enrollment/randomization, and immediately shipped to a Novartis designated central laboratory for MRD testing.
* Systemic GvHD (graft versus host disease) prophylaxis or treatment [immunosuppressive treatment (IST)] completely tapered for at least two weeks prior to study entry. Prednisone dose ≤ 5 mg/day or equivalent corticosteroid dose is allowed.
* Participants who are found with MRD positivity while still on or tapering systemic GvHD prophylaxis or treatment, MRD positivity must be re-confirmed at least 2 week after the last dose of IST
* For the adult cohorts, participants must have an Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1 or 2.

For the adolescent cohort, participants must have a Karnofsky (age ≥ 16 years) or Lansky (age < 16 years) performance status score ≥ 50%.

Exclusion Criteria:

* Prior exposure to TIM-3 directed therapy at anytime.
* History of severe hypersensitivity reactions to any ingredient of study drug(s) (azacitidine, sabatolimab) or monoclonal antibodies (mAbs) and/or their excipients
* Active Hepatitis B (HBV) or Hepatitis C (HCV) infection. Participants whose disease is controlled under antiviral therapy should not be excluded.
* Active acute GvHD grade III-IV according to standard criteria (Harris 2016).
* Active moderate chronic GvHD of the lungs according to NIH consensus criteria. Active severe chronic GvHD according to NIH consensus criteria.
* History of another primary malignancy that is currently clinically significant or currently requires active intervention. Participants who are receiving adjuvant therapy, such as hormone therapy, are eligible
* Any concurrent severe and/or active uncontrolled infection requiring parenteral antibacterial, antiviral or antifungal therapy (such as severe pneumonia, meningitis, or septicemia)
* Active autoimmune disease requiring systemic therapy (e.g. corticosteroids). Topical, inhaled, nasal and ophthalmic steroids are not prohibited. Replacement corticosteroids therapy is allowed and not considered a form of systemic treatment
* Live vaccine administered within 30 days prior to the first day of study treatment (Cycle 1 Day 1)
* Other concurrent severe and/or uncontrolled medical conditions (e.g. uncontrolled diabetes mellitus, chronic obstructive or chronic restrictive pulmonary disease including dyspnoea at rest from any cause) or history of serious organ dysfunction or disease involving the heart, kidney, or liver

Ages: 12 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2021-09-14 (Actual); Primary Completion 2024-08-22 (Actual); Study Completion 2024-08-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (9):
- Novartis Investigative Site, Marseille, France
- Germany (3):
  - Novartis Investigative Site, Freiburg im Breisgau
  - Novartis Investigative Site, Hamburg
  - Novartis Investigative Site, Münster
- Italy (4):
  - Novartis Investigative Site, Bergamo, BG
  - Novartis Investigative Site, Bologna, BO
  - Novartis Investigative Site, Brescia, BS
  - Novartis Investigative Site, Roma, RM
- Novartis Investigative Site, Barcelona, Catalonia, Spain

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent expert panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data is currently available according to the process described on www.clinicalstudydatarequest.com.
URL: http://www.clinicalstudydatarequest.com

REFERENCES:
- See also: A Plain Language Trial Summary is available on www.novctrd.com — https://www.novctrd.com/ctrdweb/patientsummary/patientsummaries?patientSummaryId=2540

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 24 participants were enrolled in this study: 21 in Safety run-in sabatolimab monotherapy and 3 in Expansion part.
Pre-assignment Details: Due to the recruitment halt by Novartis, recruitment in the expansion phase was not completed.
Groups:
- Sabatolimab 400mg Mono Adults: Safety run-in cohort: Adult participants in this arm received sabatolimab 400mg only.
- Sabatolimab 800mg Mono Adults: Safety run-in cohort: Adult participants in this arm received sabatolimab 800mg only.
- Sabatolimab 800mg + Azacitidine Adults: Expansion cohort: Adult participants in this arm received sabatolimab 800 mg + azacitidine combination
- Sabatolimab 800mg Mono Adolescent: Adolescent safety cohort: ≥12 to < 18-year-old adolescent participants in this arm received sabatolimab 800mg only.
Period: Overall Study
Arm/Group | Sabatolimab 400mg Mono Adults | Sabatolimab 800mg Mono Adults | Sabatolimab 800mg + Azacitidine Adults | Sabatolimab 800mg Mono Adolescent
Started | 10 | 11 | 2 | 1
Did Not Enter Post-treatment Follow-up (f/u) | 7 | 9 | 2 | 1
Entered Post-treatment f/u, Discontinued | 3 | 2 | 0 | 0
Completed Treatment | 2 | 0 | 0 | 0
Completed | 1 | 7 | 0 | 1
Not Completed | 9 | 4 | 2 | 0
Not completed — Death | 5 | 2 | 0 | 0
Not completed — Terminated by Sponsor | 3 | 2 | 2 | 0
Not completed — Physician Decision | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Full Analysis Set (FAS) included all participants who received at least one dose of any component of the study treatment (i.e. at least one dose of sabatolimab or at least one dose of azacitidine).
Groups:
- Total: Total of all reporting groups
Arm/Group | Sabatolimab 400mg Mono Adults | Sabatolimab 800mg Mono Adults | Sabatolimab 800mg + Azacitidine Adults | Sabatolimab 800mg Mono Adolescent | Total
Number analyzed (Participants) | 10 | 11 | 2 | 1 | 24
Age, Customized [Number; unit: Participants]
  Category 1 : 12 - <18 years | 0 | 0 | 0 | 1 | 1
  Category 1 : 18 - <65 years | 8 | 7 | 1 | 0 | 16
  Category 1 : 65 - <85 years | 2 | 4 | 1 | 0 | 7
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 6 | 2 | 1 | 14
  Male | 5 | 5 | 0 | 0 | 10
Race/Ethnicity, Customized [Number; unit: Participants]
  White | 9 | 9 | 2 | 1 | 21
  Unknown | 1 | 2 | 0 | 0 | 3

OUTCOME MEASURES:

1. Primary Outcome: Rate of Dose Limiting Toxicities (Safety Run-in in Adult Sabatolimab 400mg & 800mg Only)
Description: Assessment of tolerability of sabatolimab in adults and adolescents in the post allogenic stem cell transplantation setting. This was determined by the number of participants with at least one event - All grades. A dose-limiting toxicity (DLT) is defined as an adverse event or abnormal laboratory value considered by the Investigator to be at least possibly related to sabatolimab as a single contributor that occurs during the DLT observation period and meets the severity criteria as per protocol.
Time Frame: From Cycle 1 Day 1 to end of Cycle 2; Cycle =28 Days
Population: Dose Determining Set included all participants from the FAS enrolled in the safety run-in part who met the minimum exposure criterion described and had sufficient safety evaluations or experienced a dose limiting toxicity (DLT) between Cycle 1 Day 1 (first dose of sabatolimab) and the end of Cycle 2 (both inclusive).
Measure: Count of Participants; unit: Participants
Arm/Group | Sabatolimab 400mg Mono Adults | Sabatolimab 800mg Mono Adults
Number analyzed (Participants) | 8 | 10
Participants | 0 | 1

2. Primary Outcome: Percentage of Adult Subjects With Absence of Hematologic Relapse Per Investigator Assessment (Safety Run-in and Expansion)
Description: The percentage of adult participants for whom no evidence of hematologic relapse (no evidence of bone marrow blasts ≥5%, no evidence of reappearance of blasts in the blood; no evidence of development of extramedullary disease) has been documented after 6 cycles of study treatment or earlier discontinuation at the recommended dose of sabatolimab 800 mg.
Time Frame: From Cycle 1 Day 1 to end of Cycle 6; Cycle = 28 Days
Population: All adult participants treated with sabatolimab 800 mg monotherapy.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Sabatolimab 400mg Mono Adults | Sabatolimab 800mg Mono Adults | Sabatolimab 800mg + Azacitidine Adults | Sabatolimab 800mg Mono Adolescent
Number analyzed (Participants) | 0 | 11 | 0 | 0
Percentage of participants |  | 36.4 [10.9 to 69.2] |  |

3. Primary Outcome: Rate of Dose Limiting Toxicities (Safety Confirmation in Adolescent Cohort Only)
Description: Assessment of tolerability of sabatolimab in adolescent participants in the post allogeneic stem cell transplantation setting. This was determined by the number of participants with at least one event - All grades. A dose-limiting toxicity (DLT) is defined as an adverse event or abnormal laboratory value considered by the Investigator to be at least possibly related to sabatolimab as a single contributor that occurs during the DLT observation period and meets the severity criteria as per protocol.
Time Frame: From Cycle 1 Day 1 to end of Cycle 2; Cycle =28 Days
Population: Dose Determining Set included all participants from the FAS enrolled in the adolescent cohort who met the minimum exposure criterion described and had sufficient safety evaluations or experienced a dose limiting toxicity (DLT) between Cycle 1 Day 1 (first dose of sabatolimab) and the end of Cycle 2 (both inclusive).
Measure: Count of Participants; unit: Participants
Arm/Group | Sabatolimab 800mg Mono Adolescent
Number analyzed (Participants) | 1
Participants | 0

4. Secondary Outcome: Incidence of Grade III or IV Acute Graft Versus Host Disease (aGvHD)
Description: Assessment of the treatment emergent grade III or IV aGvHD. Acute GvHD: Grade IV acute GvHD, Stage ≥3 lower GI acute GvHD (consistent with Grade III acute GvHD) or Stage ≥3 liver acute GvHD (consistent with Grade III GvHD).
Time Frame: From start of treatment to up to 36 months from last patient first treatment.
Population: Safety Set includes all participants from the FAS.
Measure: Number; unit: Participants
Arm/Group | Sabatolimab 400mg Mono Adults | Sabatolimab 800mg Mono Adults | Sabatolimab 800mg + Azacitidine Adults | Sabatolimab 800mg Mono Adolescent
Number analyzed (Participants) | 10 | 11 | 2 | 1
Participants | 0 | 0 | 0 | 0

5. Secondary Outcome: Incidence of Moderate to Severe Chronic GVHD (cGvHD)
Description: Assessment of the treatment emergent moderate or severe cGvHD. Chronic GvHD: Moderate chronic GvHD of the lungs, Severe chronic GvHD.
Time Frame: From start of treatment to up to 36 months from last patient first treatment.
Population: Safety Set includes all participants from the FAS.
Measure: Count of Participants; unit: Participants
Arm/Group | Sabatolimab 400mg Mono Adults | Sabatolimab 800mg Mono Adults | Sabatolimab 800mg + Azacitidine Adults | Sabatolimab 800mg Mono Adolescent
Number analyzed (Participants) | 10 | 11 | 2 | 1
Participants | 0 | 1 | 0 | 0

6. Secondary Outcome: Peak of Serum Concentration (Cmax) Sabatolimab
Description: Cmax is the maximal serum concentration of sabatolimab.
Time Frame: Cycle 1 Day 5 (end of infusion) and Cycle 3 Day 1 or Day 5 (end of infusion) and Cycle 24 Day 1 (end of infusion); Cycle =28 Days
Population: Pharmacokinetics (PK) analysis set included all participants from the Safety Set who provided at least one evaluable sabatolimab PK concentration at the considered timepoint.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ug/ml
Arm/Group | Sabatolimab 400mg Mono Adults | Sabatolimab 800mg Mono Adults | Sabatolimab 800mg + Azacitidine Adults | Sabatolimab 800mg Mono Adolescent
Number analyzed (Participants) | 6 | 7 | 1 | 0
ug/ml
  Cycle 1 Day 5 at 2 hours (hr) (end of infusion): number analyzed (Participants) | 0 | 0 | 1 | 0
  Cycle 1 Day 5 at 2 hours (hr) (end of infusion) |  |  | 256 (0.0) |
  Cycle 3 Day 1 at 2 hr (end of infusion): number analyzed (Participants) | 6 | 7 | 0 | 0
  Cycle 3 Day 1 at 2 hr (end of infusion) | 137 (52.7) | 304 (31.4) |  |
  Cycle 3 Day 5 at 2 hr (end of infusion): number analyzed (Participants) | 0 | 0 | 1 | 0
  Cycle 3 Day 5 at 2 hr (end of infusion) |  |  | 315 (0.0) |
  Cycle 24 Day 1 at 2 hr (end of infusion): number analyzed (Participants) | 2 | 0 | 0 | 0
  Cycle 24 Day 1 at 2 hr (end of infusion) | 163 (23.7) |  |  |

7. Secondary Outcome: Trough Serum Concentration of (Cmin) Sabatolimab
Description: Cmin is the concentration of sabatolimab prior to next dosing or after end of treatment.
Time Frame: Adult cohorts: Pre-dose on Day 1 (safety run-in) or Day 5 (expansion) of Cycle 1, 3, 6 and 24 (safety run-in only); Adolescent cohort: Pre-dose on Day 1 of Cycle 1, 2, 3 and 6; Cycle = 28 Days
Population: as for outcome 6
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µg/ml
Arm/Group | Sabatolimab 400mg Mono Adults | Sabatolimab 800mg Mono Adults | Sabatolimab 800mg + Azacitidine Adults | Sabatolimab 800mg Mono Adolescent
Number analyzed (Participants) | 6 | 7 | 2 | 1
µg/ml
  0-hour (hr) Pre-dose at Cycle 1 Day 1: number analyzed (Participants) | 6 | 7 | 0 | 1
  0-hour (hr) Pre-dose at Cycle 1 Day 1 | 0.00 (0.0) | 0.00 (0.0) |  | 0.00 (0.0)
  0 hr (pre-dose) at Cycle 1 Day 5: number analyzed (Participants) | 0 | 0 | 2 | 0
  0 hr (pre-dose) at Cycle 1 Day 5 |  |  | 0.00 (0.0) |
  0 hr (pre-dose) at Cycle 2 Day 1: number analyzed (Participants) | 0 | 0 | 0 | 1
  0 hr (pre-dose) at Cycle 2 Day 1 |  |  |  | 70.7 (0.0)
  0 hr (pre-dose) at Cycle 3 Day 1: number analyzed (Participants) | 6 | 7 | 0 | 1
  0 hr (pre-dose) at Cycle 3 Day 1 | 40.4 (20.2) | 70.7 (47.5) |  | 129 (0.0)
  0 hr (pre-dose) at Cycle 3 Day 5: number analyzed (Participants) | 0 | 0 | 1 | 0
  0 hr (pre-dose) at Cycle 3 Day 5 |  |  | 42.9 (0.0) |
  0 hr (pre-dose) at Cycle 6 Day 1: number analyzed (Participants) | 4 | 5 | 0 | 1
  0 hr (pre-dose) at Cycle 6 Day 1 | 46.4 (66.4) | 99.8 (52.1) |  | 219 (0.0)
  0 hr (pre-dose) at Cycle 6 Day 5: number analyzed (Participants) | 0 | 0 | 1 | 0
  0 hr (pre-dose) at Cycle 6 Day 5 |  |  | 71.9 (0.0) |
  0 hr (pre-dose) at Cycle 24 Day 1: number analyzed (Participants) | 2 | 0 | 0 | 0
  0 hr (pre-dose) at Cycle 24 Day 1 | 49.7 (44.1) |  |  |

8. Secondary Outcome: Graft Versus Host Disease (GvHD)-Free/Relapse-free Survival (GRFS)
Description: Time from start of treatment to the date of first documented occurrence or worsening of treatment emergent grade III or IV aGvHD or moderate to severe cGvHD requiring initiation of systemic treatment, morphologic/hematologic relapse, or death due to any cause, whichever occurs first
Time Frame: From start of treatment to up to 36 months from last patient first treatment
Population: as for baseline characteristics
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Sabatolimab 400mg Mono Adults | Sabatolimab 800mg Mono Adults | Sabatolimab 800mg + Azacitidine Adults | Sabatolimab 800mg Mono Adolescent
Number analyzed (Participants) | 10 | 11 | 2 | 1
Months | NA [NA to NA] — NA: Not estimable due to insufficient number of participants with events resulting from the early termination of the study in part 2 (expansion cohort). | NA [NA to NA] — NA: Not estimable due to insufficient number of participants with events resulting from the early termination of the study in part 2 (expansion cohort). | NA [NA to NA] — NA: Not estimable due to insufficient number of participants with events resulting from the early termination of the study in part 2 (expansion cohort). | NA [NA to NA] — NA: Not estimable due to insufficient number of participants with events resulting from the early termination of the study in part 2 (expansion cohort).

9. Secondary Outcome: Relapse-free Survival (RFS)
Description: Time from start of treatment to the date of first documented hematologic relapse or death due to any cause, whichever occurs first.
Time Frame: From start of treatment to up to 36 months from last patient first treatment
Population: FAS included all participants who received at least one dose of any component of the study treatment (i.e. at least one dose of sabatolimab or at least one dose of azacitidine).
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Sabatolimab 400mg Mono Adults | Sabatolimab 800mg Mono Adults | Sabatolimab 800mg + Azacitidine Adults | Sabatolimab 800mg Mono Adolescent
Number analyzed (Participants) | 10 | 11 | 2 | 1
Months | 2.56 [0.95 to NA] — NA: The upper limit of Confidence Interval (CI) was not estimable due to an insufficient number of participants and limited follow-up, resulting from the early termination of the study in part 2 (expansion cohort). | 6.74 [0.95 to NA] — NA: The upper limit of CI was not estimable due to an insufficient number of participants and limited follow-up, resulting from the early termination of the study in part 2 (expansion cohort). | NA [NA to NA] — NA: CI was not estimable as no participants had an event within the limited number of participants, resulting from the early termination of the study in part 2 (expansion cohort). | 7.16 [NA to NA] — NA: The CI was not estimable due to the limited number of participants, resulting from the early termination of the study in part 2 (expansion cohort).

10. Secondary Outcome: Percentage of Participants With Measurable Residual Disease (MRD) Positive at Baseline Who Become MRD Negative
Description: Percentage of participants with centrally confirmed MRD+ status at baseline converting to MRD- within the first 6 cycles of study treatment.
Time Frame: From start of treatment until end of Cycle 6 (Cycle = 28 Days)
Population: as for outcome 9
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Sabatolimab 400mg Mono Adults | Sabatolimab 800mg Mono Adults | Sabatolimab 800mg + Azacitidine Adults | Sabatolimab 800mg Mono Adolescent
Number analyzed (Participants) | 10 | 11 | 2 | 1
Percentage of participants | 0 [0.0 to 30.8] | 0 [0.0 to 28.5] | 0 [0.0 to 84.2] | 0 [0.0 to 97.5]

ADVERSE EVENTS:
Time Frame: Adverse Events were collected from start of treatment (FPFT) up to 30 days after the last dose of study treatment (sabatolimab or azacitidine), for a maximum duration of approx. 25 months (max. duration of treatment 24 months + 30 days). Deaths were collected on-treatment period up to 30 days and after Day 31 after last dose of study treatment.
Description: An Adverse Event is any sign or symptom occurring during a trial and safety follow-up. The Safety Set comprises all participants who received at least one dose of any component of the study treatment (i.e. at least one dose of sabatolimab or at least one dose of azacitidine).
Arm/Group | Sabatolimab 400mg Mono Adults | Sabatolimab 800mg Mono Adults | Sabatolimab 800mg + Azacitidine Adults | Sabatolimab 800mg Mono Adolescent
All-Cause Mortality (participants affected / at risk) | 5/10 | 2/11 | 0/2 | 0/1
Serious Adverse Events (participants affected / at risk) | 2/10 | 3/11 | 0/2 | 0/1
Other Adverse Events (participants affected / at risk) | 9/10 | 9/11 | 2/2 | 1/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sabatolimab 400mg Mono Adults (N=10) | Sabatolimab 800mg Mono Adults (N=11) | Sabatolimab 800mg + Azacitidine Adults (N=2) | Sabatolimab 800mg Mono Adolescent (N=1)
Myocarditis (Cardiac disorders) | 0 | 1 | 0 | 0
Bronchitis (Infections and infestations) | 1 | 0 | 0 | 0
Febrile infection (Infections and infestations) | 1 | 0 | 0 | 0
Oral herpes (Infections and infestations) | 0 | 1 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 0 | 0
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Nervous system disorder (Nervous system disorders) | 0 | 1 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Sabatolimab 400mg Mono Adults (N=10) | Sabatolimab 800mg Mono Adults (N=11) | Sabatolimab 800mg + Azacitidine Adults (N=2) | Sabatolimab 800mg Mono Adolescent (N=1)
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 2 | 1 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 3 | 0 | 0 | 0
Tachycardia (Cardiac disorders) | 0 | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 1 | 2 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Asthenia (General disorders) | 1 | 1 | 1 | 0
Chest pain (General disorders) | 1 | 0 | 0 | 0
Fatigue (General disorders) | 1 | 1 | 1 | 0
Influenza like illness (General disorders) | 0 | 1 | 0 | 0
Injection site pain (General disorders) | 0 | 0 | 1 | 0
Mucosal inflammation (General disorders) | 0 | 1 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 0 | 1 | 0
Oedema (General disorders) | 1 | 0 | 0 | 0
Oedema peripheral (General disorders) | 0 | 1 | 0 | 0
Pyrexia (General disorders) | 0 | 1 | 0 | 0
Chronic graft versus host disease (Immune system disorders) | 0 | 1 | 0 | 0
Bronchitis (Infections and infestations) | 1 | 0 | 0 | 0
COVID-19 (Infections and infestations) | 2 | 2 | 1 | 1
Clostridium difficile colitis (Infections and infestations) | 1 | 0 | 0 | 0
Febrile infection (Infections and infestations) | 0 | 1 | 0 | 0
Folliculitis (Infections and infestations) | 1 | 0 | 0 | 0
Herpes zoster (Infections and infestations) | 1 | 0 | 0 | 0
Influenza (Infections and infestations) | 0 | 1 | 0 | 0
Metapneumovirus infection (Infections and infestations) | 1 | 0 | 0 | 0
Oral bacterial infection (Infections and infestations) | 0 | 0 | 1 | 0
Oral candidiasis (Infections and infestations) | 0 | 0 | 1 | 0
Otitis media (Infections and infestations) | 1 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 0 | 0
Rhinitis (Infections and infestations) | 0 | 0 | 1 | 1
Viral infection (Infections and infestations) | 0 | 1 | 0 | 0
Anaemia postoperative (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Immunisation reaction (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 1 | 1 | 1 | 0
Amylase increased (Investigations) | 1 | 0 | 1 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 1 | 1 | 0
Blood alkaline phosphatase increased (Investigations) | 1 | 1 | 1 | 0
Blood cholesterol increased (Investigations) | 0 | 1 | 0 | 0
Blood creatinine increased (Investigations) | 0 | 1 | 0 | 0
Blood potassium increased (Investigations) | 0 | 0 | 1 | 0
Brain natriuretic peptide increased (Investigations) | 1 | 0 | 0 | 0
C-reactive protein increased (Investigations) | 1 | 0 | 0 | 0
Gamma-glutamyltransferase increased (Investigations) | 1 | 1 | 1 | 0
Lipase increased (Investigations) | 1 | 0 | 1 | 0
Troponin T increased (Investigations) | 0 | 1 | 0 | 0
White blood cell count increased (Investigations) | 0 | 0 | 1 | 0
Cachexia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Hyperferritinaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Tumour lysis syndrome (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Neuropathy peripheral (Nervous system disorders) | 1 | 0 | 0 | 0
Paraesthesia (Nervous system disorders) | 0 | 0 | 1 | 0
Somnolence (Nervous system disorders) | 0 | 0 | 1 | 0
Dysuria (Renal and urinary disorders) | 1 | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 0 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Intertrigo (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Telangiectasia (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Hypertensive crisis (Vascular disorders) | 0 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of pooled data (i.e.,data from all sites) in clinical trial or disclosure of trial results in their entirety.

DOCUMENTS (2):
  • Study Protocol (2022-03-24): https://cdn.clinicaltrials.gov/large-docs/16/NCT04623216/Prot_000.pdf
  • Statistical Analysis Plan (2024-07-03): https://cdn.clinicaltrials.gov/large-docs/16/NCT04623216/SAP_001.pdf